CLINICAL TRIAL: NCT00464061
Title: Efficacy and Safety of 2mg/Day of M100907 on Sleep Maintenance Insomnia With a Sub-study of the Effect of M100907 on Stable Type II Diabetes Mellitus: a One Year, Multi-center, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy an Safety of Volinanserin on Sleep Maintenance Insomnia With a Sub-study on Stable Type II Diabetes Mellitus
Acronym: SAMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision due to absence of demonstration of efficacy of volinanserin in primary insomnia with predominant sleep maintenance problems
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTE6673; EudraCT : 2006-004942-18
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep problems; Insomnia; Sleeplessness; Primary insomnia; Insomnia disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — volinanserin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Volinanserin (Experimental)
  Interventions: Drug: Volinanserin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Volinanserin — oral administration
  Other Names: M100907
  Arms: Volinanserin
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess efficacy and safety of volinanserin in the population of patients complaining of sleep maintenance insomnia. The objective of the substudy is to assess glycemic control in the subgroup of patients with type II diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on Diagnostic and Statistical Manual of Mental Disorders (Fourth Edition) criteria
* Disturbances of sleep maintenance criteria based on participant's information related to sleep pattern during the preceding month

Sub-study :

* Participants will be included if they have an established medical diagnosis of type II Diabetes Mellitus, and have been treated either with an oral hypoglycemic agent and/or insulin for at least three months prior to the Screening Visit (with stable regimen for at least one month prior to screening)

Exclusion Criteria:

* Females who are lactating or who are pregnant
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month
* Consumption of xanthine-containing beverages (i.e. tea, coffee, cola) comprising more than 5 cups/day
* Participation in another trial having received study medication within 1 month before the screening visit
* Body Mass Index ≥ 33
* Use of over-the-counter medications such as tryptophan, valerian root, kava, melatonin, St. John's Wort, Alluna or prescription sleep medication
* Use of any substance with psychotropic effects or properties know to affect sleep/wake
* History of primary hypersomnia, narcolepsy, breathing-related sleep disorder, circadian rhythm sleep disorder, parasomnia, dyssomnia
* Clinically significant, severe or unstable, acute or chronically progressive medical or surgical disorder
* Positive qualitative urine drug screen (opiates, cocaine, amphetamine…)

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1847 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: change from baseline for Sleep Maintenance Insomnia using patient reported Wake After Sleep Onset (pr-WASO) | at 3 months
Efficacy (sub-study): change from baseline for glycemic measure HbA1c | at 6 and 12 months

SECONDARY OUTCOMES:
Efficacy: change from baseline of the pr-WASO | at 6 and 12 months
Efficacy: change from baseline of "General Productivity" domain score of the Functional Outcomes of Sleep Questionnaire | at 3 months
Safety: adverse events and laboratory abnormalities | during 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (22):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Anofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom